CLINICAL TRIAL: NCT07037147
Title: To Compare the Efficacy of Instrument Assisted Soft Tissue Mobilization vs Bowen Therapy in Alleviating Pain and Tightness of Trapezius Muscle
Brief Title: To Compare the Efficacy of Instrument Assisted STM vs BT in Alleviating Pain and Tightness of Trapezius Muscle
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall20/1007
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Trapezius Muscle Strain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- instrument assistance soft tissue mobilisation (Experimental)
  Interventions: Combination Product: instrument assistance soft tissue mobilisation
- Bowen technique (Experimental)
  Interventions: Combination Product: Bowen technique

INTERVENTIONS:
Combination Product: instrument assistance soft tissue mobilisation — In this group instrument assistance soft tissue mobilisation will be given followed by conventional therapy. IASTM will be given by using IASTM tool M2T blade. In this process patient will be asked to sit in a chair by resting its forearm in front of the table.
  Arms: instrument assistance soft tissue mobilisation
Combination Product: Bowen technique — In this group Bowen technique will be given after the basic conventional therapy. For this technique patient will be asked to lie in a prone position where the neck of the patient will be supported with the help of a small pillow. Therapist thumb will be placed on the affected side of the muscle.
  Arms: Bowen technique

SUMMARY:
Trapezius muscle pain and tightness are common musculoskeletal issues that can significantly impair movement and quality of life. Instrument Assisted Soft Tissue Mobilization (IASTM) and Bowen Therapy are gaining attention as non-invasive treatments for myofascial pain and tension.

DETAILED DESCRIPTION:
It will be single blinded randomized clinical trial (RCT). The study will be conducted on 26 participants which will be categorized into two groups. Group one will be given IASTM and group two will receive Bowen technique. Non-probability convenience sampling technique will be used for data collection at physiotherapy department at Fatima memorial hospital followed by lottery method of allocation of groups. Data will be collected by using visual analogue scale, goniometer and neck disability index.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 50 years
* Both gender
* Bilateral trapezius muscle tightness assessed by palpation.
* Subject with the presence of myofacial trigger points in upper trapezius muscle assessed on palpation.
* Patient with symptoms for the past two weeks.
* People with pain of neck due to tight muscle more than 3 on VAS.

Exclusion Criteria:

* Participant with any fracture of cervical spine or surgery within the 6 month timespan.
* Participant with radiating neck pain towards the upper extremity.
* People with other conditions like disc prolapse, spondylolisthesis, tb of spine etc.
* People with any instrument assistance soft tissue mobilisation technique contraindication.
* People with whiplash injury history.
* Participant who has been diagnosed with myopathy or fibromyalgia.
* Pregnant females who has already gone under myofacial therapy within the past month.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | 6 Months
  Visual analogue scale is known pain assessment scale which was introduced by Hayes and Patterson in 1921. Its scoring range is from 0 to 10 where 0 shows no pain, 5 shows moderate pain and 10 shows worst pain.
Neck Disability Index | 6 Months
  Neck pain disability index is used for the disability of the neck or the impact of neck pain on a person. This 10 item questionnaire is used to assess the patient overall quality of life as well as the personal ability to perform activities of daily living.
Neck Disability Index | 6 months
  Neck disability index is used for the disability of the neck or the impact of neck pain on a person. This 10 item questionnaire is used to assess the patient overall quality of life as well as the personal ability to perform activities of daily living.

CONTACTS AND LOCATIONS:
Locations (1):
- Fatima Memorial Hospital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No